CLINICAL TRIAL: NCT03420911
Title: Determination of the Effects of Change in Anxiety Level on Pain Perception in Patients Who Present to Emergency Department Due to Acute Pain: a Double Blind, Randomized, Controlled Trial
Brief Title: Determination of the Effects of Change in Anxiety Level on Pain Perception in Patients Who Present to Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ASIM ENES ÖZBEK, Principal Investigator, Derince Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013/147
Record Dates: First submitted 2018-01-16; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Pain, Acute; Anxiety
Keywords: pain; anxiety; emergency department; pain management
MeSH Terms: conditions — Acute Pain; Anxiety Disorders; Pain; Emergencies; Agnosia | interventions — dexketoprofen trometamol; Midazolam

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned into two groups with a 1:1 allocation following simple randomization procedures by a program generating an online random number
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sequenced study medications were prepared by a nurse, and another nurse administered the medications.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexketoprofen trometamol group (Active Comparator): Received the study drugs in 100 mL of normal saline within 5 minutes. The dexketoprofen trometamol dose was 50 mg
  Interventions: Drug: dexketoprofen trometamol
- dexketoprofen trometamol plus midazolam group (Active Comparator): Received the study drugs in 100 mL of normal saline within 5 minutes. The dexketoprofen trometamol dose was 50 mg and the midazolam dose was 1 mg.
  Interventions: Drug: dexketoprofen trometamol; Drug: Midazolam

INTERVENTIONS:
Drug: dexketoprofen trometamol
Drug: Midazolam
  Arms: dexketoprofen trometamol plus midazolam group

SUMMARY:
The aim of this study is to determine the level of pain and anxiety in patients who present to the emergency department with acute pain, and to investigate the effect of the standard analgesic treatment and an additional anxiolytic treatment on pain and anxiety.

DETAILED DESCRIPTION:
After triage, each acute pain patient who qualified for the study was asked for consent. Written informed consent was obtained from all patients who were eligible for the study. After obtaining written informed consent, demographic and clinical data were collected and recorded by the attending physician. Our study consisted of two parallel groups. Participants were randomly assigned into two groups with a 1:1 allocation following simple randomization procedures by a program generating an online random number. The control group was given only the analgesic drug dexketoprofen trometamol and the study group was given analgesic plus anxiolytic, the same dose of dexketoprofen trometamol plus midazolam . Both groups received the study drugs in 100 mL of normal saline within 5 minutes. The dexketoprofen trometamol dose was 50 mg, and the midazolam dose was 1 mg. The study was double-blind. Sequenced study medications were prepared by a nurse, and another nurse administered the medications. In patients with an insufficient improvement of pain after 60 minutes, fentanyl 1 mcg/kg ı.v. was administered as a rescue medication.

Pain and anxiety in patients was measured at 0, 30, 60 and 120 minutes using the standard 100 mm horizontal visual analogue scale (VAS). The patient's general anxiety states were measured with the Turkish adopted version of the Hospital Anxiety and Depression Scale (HADS). Patients who have greater than 10 points are assumed anxious (9). The HADS and VAS scores were measured and recorded to the database by the researcher. At the time of discharge, patient satisfaction with treatment was evaluated by asking two questions with the 5-step Likert scale. The questions were, "I am satisfied with the applied treatment", and "I would like the same treatment applied again". Patient answers were, "1-I strongly disagree", "2-I disagree", "3-I am not sure", "4-I agree", and "5-I strongly agree".

ELIGIBILITY:
Inclusion Criteria:

* The patients who presented to the emergency department with acute pain
* Who accepted to include the study
* Who were older than 18 years old

Exclusion Criteria:

* Patients who refused to participate to the study
* History of allergy to any of the study drugs
* Pregnancy
* Younger than 18 years old
* Chronic pain
* Antidepressant or anxiolytic drug use
* Advanced kidney or liver failure
* Use of analgesics within 6 hours before presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
the change in pain levels | 30 minutes
  the change in pain levels between groups on the 100mm visual analogue scale at 0-30th minutes
the change in anxiety levels | 30 minutes
  the change in anxiety levels between groups on the 100mm visual analogue scale at 0-30th minutes

SECONDARY OUTCOMES:
the need for rescue treatment | 120 minutes
  the need for rescue treatment at 60th minute and at 120 th minute
the rate of the request for the same treatment | 120 minutes
  the rate of the request for the same treatment again on the Likert scale
the comparison of the pain and anxiety change on the visual analogue scale | 120 minutes
  the comparison of the pain and anxiety change on the visual analogue scale in patients who have a greater anxiety score.

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Tanabe P, Buschmann M. A prospective study of ED pain management practices and the patient's perspective. J Emerg Nurs. 1999 Jun;25(3):171-7. doi: 10.1016/s0099-1767(99)70200-x. PMID 10346837
- [Background] Karwowski-Soulie F, Lessenot-Tcherny S, Lamarche-Vadel A, Bineau S, Ginsburg C, Meyniard O, Mendoza B, Fodella P, Vidal-Trecan G, Brunet F. Pain in an emergency department: an audit. Eur J Emerg Med. 2006 Aug;13(4):218-24. doi: 10.1097/01.mej.0000217975.31342.13. PMID 16816586
- [Background] Craven P, Cinar O, Madsen T. Patient anxiety may influence the efficacy of ED pain management. Am J Emerg Med. 2013 Feb;31(2):313-8. doi: 10.1016/j.ajem.2012.08.009. Epub 2012 Sep 13. PMID 22981626
- [Background] Ocanez KL, McHugh RK, Otto MW. A meta-analytic review of the association between anxiety sensitivity and pain. Depress Anxiety. 2010 Aug;27(8):760-7. doi: 10.1002/da.20681. PMID 20336798
- [Background] Ethier C, Burry L, Martinez-Motta C, Tirgari S, Jiang D, McDonald E, Granton J, Cook D, Mehta S; Canadian Critical Care Trials Group. Recall of intensive care unit stay in patients managed with a sedation protocol or a sedation protocol with daily sedative interruption: a pilot study. J Crit Care. 2011 Apr;26(2):127-32. doi: 10.1016/j.jcrc.2010.08.003. PMID 20889289
- [Background] Behrbalk E, Halpern P, Boszczyk BM, Parks RM, Chechik O, Rosen N, Shapira A, Merose O, Uri O. Anxiolytic medication as an adjunct to morphine analgesia for acute low back pain management in the emergency department: a prospective randomized trial. Spine (Phila Pa 1976). 2014 Jan 1;39(1):17-22. doi: 10.1097/BRS.0000000000000038. PMID 24270933
- [Background] Bonett DG, Price RM. Statistical inference for a linear function of medians: confidence intervals, hypothesis testing, and sample size requirements. Psychol Methods. 2002 Sep;7(3):370-83. doi: 10.1037/1082-989x.7.3.370. PMID 12243307
- [Background] Mok LC, Lee IF. Anxiety, depression and pain intensity in patients with low back pain who are admitted to acute care hospitals. J Clin Nurs. 2008 Jun;17(11):1471-80. doi: 10.1111/j.1365-2702.2007.02037.x. Epub 2008 Feb 19. PMID 18298508
- [Background] Oktay C, Eken C, Ozbek K, Ankun G, Eray O, Avci AB. Pain perception of patients predisposed to anxiety and depressive disorders in emergency department. Pain Manag Nurs. 2008 Dec;9(4):150-3, 153.e1-3. doi: 10.1016/j.pmn.2008.06.002. PMID 19041612
- See also: Pain clinical manual / Margo McCaffery, Chris Pasero. — http://www.ncbi.nlm.nih.gov/nlmcatalog/100889125
- See also: IASP Task Force on Taxonomy Part III: Pain Terms, A Current List with Definitions and Notes on Usage. IASP Task Force Taxon. — http://www.iasp-pain.org/Taxonomy